CLINICAL TRIAL: NCT02710552
Title: Randomized Comparison of Fixed Low-dose Combination of THREE Antihypertensive Drugs Versus Fixed High-dose Combination of Two Antihypertensive Drugs in Arterial Hypertension (the 3D Trial)
Brief Title: Low-dose Combination of Three Antihypertensive Drugs
Acronym: 3D
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123/D/2016
Record Dates: First submitted 2016-03-04; First posted 2016-03-16 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Arterial Hypertension
Keywords: arterial hypertension; antihypertensive drugs
MeSH Terms: conditions — Hypertension | interventions — Perindopril; Indapamide; Amlodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Three antihypertensive Drugs (Active Comparator): Patients will be treated with Tripliam, that is a commercially available fixed low-dose combination of three antihypertensive drugs, that is 5 mg/daily perindopril, 1,25 mg/daily indapamide and 5 mg/day amlodipine
  Interventions: Drug: Tripliam (perindopril, indapamide, amlodipine)
- Two antihypertensive drugs (Active Comparator): Patients will be treated with Reaptan, that is a commercially available fixed high-dose combination of two antihypertensive drugs, that is 10 mg/daily perindopril and 5 mg/day amlodipine
  Interventions: Drug: Reaptan (perindopril, amlodipine)

INTERVENTIONS:
Drug: Tripliam (perindopril, indapamide, amlodipine) — Fixed combination of perindopril 5 mg, indapamide 1,25 and amlodipine 5 mg
  Other Names: Combination of three antihypertensive drugs
  Arms: Three antihypertensive Drugs
Drug: Reaptan (perindopril, amlodipine) — Fixed combination of perindopril 10 mg and amlodipine 5 mg
  Other Names: Combination of two antihypertensive drugs
  Arms: Two antihypertensive drugs

SUMMARY:
The aim of the study is to compare the efficacy and safety of low-dose combination of three antihypertensive drugs versus fixed high-dose combination of two antihypertensive drugs in arterial hypertension

DETAILED DESCRIPTION:
The aim of the study is to compare the efficacy and safety of commercially available low-dose combination of three antihypertensive drugs versus commercially available fixed high-dose combination of two antihypertensive drugs in arterial hypertension

ELIGIBILITY:
Inclusion Criteria:

Patients with arterial hypertension resistant to monotherapy

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients who reach target blood pressure | From baseline to the end of the 3-month study period
  How many patients have blood pressure within normal limits

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gaudio, MD, Study Chair — Sapienza University
Locations (1):
- Sapienza University, Rome, Italy

IPD SHARING:
Plan to Share IPD: No